CLINICAL TRIAL: NCT04764071
Title: Safety And Efficacy Of Ultra-Mini Percutaneous Nephrolithotomy In Comparison With Standard Percutaneous Nephrolithotomy For Management Of Renal Calyceal Calculi 1 Cm To 2 Cm In Size. Comparative Randomized Prospective Study
Brief Title: Ultra-Mini Versus Standard Percutaneous Nephrolithotomy For Management Of Renal Calculi. A Randomized Controlled Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD 06 /2020
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Intervention Model Description: To compare the difference between the two procedures regarding stone-free rates, operative time, hospital stay, procedures cost, and operative complications including blood loss, the need for blood transfusion, and extravasation or urine leakage
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, the Data Collector, and the statistician were blinded to the arms of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous nephrolithotomy (Active Comparator): Patients are positioned in the lithotomy position and a 6F ureteral catheter is placed and the bladder is drained with a 16F urethral Foley catheter. After ureteral catheterization, patients are placed in the prone position, and percutaneous access of the desired calyx is achieved under fluoroscopic guidance with the use of an 18-gauge needle and a guidewire passage. Tract dilation is accomplished by using Amplatz dilators up to 30F. Pneumatic lithotripter is used for fragmentation and stone removal is accomplished with retrieval graspers through a rigid 22F nephroscope. An 18-24 F nephrostomy tube is placed at the end of the operation.
  Interventions: Procedure: percutaneous nephrolithotomy
- ultra-mini percutaneous nephrolithotomy (Experimental): Patients are positioned in the lithotomy position and a 6 F ureteral catheter is placed and the bladder is drained with a 16F urethral Foley catheter. After ureteral catheterization, patients are placed in the prone position, and percutaneous access of the desired calyx is achieved under fluoroscopic guidance with the use of an 18-gauge needle and a guidewire passage. Tract dilation is accomplished by using Amplatz dilators up to 12-14 F fascial dilator was used to dilate the nephrostomy tract to pass the 13 F semi-rigid plastic sheath. Then, a 9.5-F, rigid ureteroscope (KARL STORZ Medical Instruments) was introduced to the sheath. The renal stones were broken into pieces using holmium laser lithotripsy. Finally, the ureteroscope and sheath were removed and the tract site was packed for 2-3 min. then placement of double J stent will be done according to the decision of the operating surgeon for 3 to 4 weeks.
  Interventions: Procedure: ultra-mini percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: percutaneous nephrolithotomy — percutaneous access of the desired calyx is achieved under fluoroscopic guidance with the use of an 18-gauge needle and a guidewire passage. Tract dilation is accomplished by using Amplatz dilators up to 30F.
  Arms: percutaneous nephrolithotomy
Procedure: ultra-mini percutaneous nephrolithotomy — percutaneous access of the desired calyx is achieved under fluoroscopic guidance with the use of an 18-gauge needle and a guidewire passage. Tract dilation is accomplished by using Amplatz dilators up to 12-14 F fascial dilator was used to dilate the nephrostomy tract to pass the 13 F semi-rigid plastic sheath.
  Arms: ultra-mini percutaneous nephrolithotomy

SUMMARY:
Renal stones are one of the most common urological problems and there are multiple methods for their management such as percutaneous nephrolithotomy, mini and ultra-mini percutaneous nephrolithotomy, flexible ureteroscopy and laser lithotripsy, and extracorporeal shock wave lithotripsy. percutaneous nephrolithotomy is the treatment of choice for the management of renal calculi, in spite of the increasing stone clearance rate, the complication rate of this procedure is relatively higher.

DETAILED DESCRIPTION:
Nephrolithiasis is a major worldwide source of morbidity, constituting a common urological disease affecting 10-15% of the world population. Consistent technical advancements provide surgeons and patients with several options for the treatment of renal calculi, including extracorporeal shock wave lithotripsy (ESWL), percutaneous nephrolithotomy (PCNL), retrograde intrarenal surgery (RIRS), and conventional open surgery.

Percutaneous nephrolithotomy (PCNL) is generally considered a gold standard in renal stones particularly larger than 2cm or lower calyceal larger than 1cm offering high stone-free rates after the first treatment as compared to the other minimal invasive lithotripsy techniques.

Percutaneous nephrolithotripsy (PCNL)is a procedure to remove kidney stones from the kidney through a small incision in the skin and it was initially described in the literature by Fernström and Johansson in 1976. Traditionally, the prone position was considered the only position to obtain renal access for PCNL. In 1987, Valdivia Urìa presented the supine PCNL.

PCNL is also recommended in the case of smaller stones in patients with contraindications for shockwave lithotripsy (SWL), such as shockwave resistant stones and anatomical malformations, or when a patient elects PCNL as a procedure of higher efficacy. However, serious complications although rare should be expected following this percutaneous procedure as, Perioperative bleeding, urine leakage from nephrocutaneous tract, pelvicalyceal system injury, pain.( Kyriazis et al 2015) colon injury, hydrothorax, pneumothorax, prolonged leak, sepsis, ureteral stone, vascular injury and acute loss of kidney, all are individually confronted complications after PCNL.

PCNL techniques include: standard PCNL (S-PCNL), mini-PCNL (also called miniperc), ultra-mini-PCNL (UM-PCNL) and the recently introduced micro-PCNL. One of the most important differences between the various PCNL techniques is the size of renal access, which contributes to the broad spectrum of complications and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patient aged over 18 with renal stone between 1 and 2 cm

Exclusion Criteria:

1. patient with a single kidney.
2. Renal stones larger than 2 cm or less than 1 cm.
3. Patients with uncontrolled co-morbidities (hypertension, diabetes mellitus, cardiac disease, chest disease).
4. Patients with active urinary tract infection.
5. Patients with other anatomic renal abnormalities (congenital renal malformations such as horseshoe kidney, polycystic kidney disease, etc.). and Patients with severe skeletal deformity.
6. Pregnant women.
7. Patients with Uncorrectable bleeding disorder.
8. Patients who underwent renal transplantation or urinary diversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-28 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
stone free rate of patients with renal stones by non contrast CT scan | first day postoperative
  efficacy of the procedure to clear renal stones completely in single session, non contrast CT will evaluate the stone burden and compare it to the preoperative measurement

SECONDARY OUTCOMES:
operative time of both procedures | intraoperative finding
  time of each procedure in minutes from the lithotomy positioning till completion of the procedure
hospital stay of the patient | 1 to 3 days postoperative
  duration till patient is discharged in days
hemoglobin drop of the patients | first day postoperative
  decrease in the hemoglobin level in comparison to the preoperative results
postoperative urine leakage from the surgical wound | first day postoperative
  urine leakage from the nephrostomy site if it present or not as document during surgical dressing by the attending physician
cost analysis of both procedure | 3 days postoperative
  cost of each procedure including operative cost and postoperative stay in Egyptian Pound

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
To compare the difference between the two procedures regarding stone-free rates, operative time, hospital stay, procedures cost, and operative complications including blood loss, the need for blood transfusion, and extravasation or urine leakage.